CLINICAL TRIAL: NCT05589662
Title: Analysis of Clinical, Functional and Musculoskeletal Variables Between Adult Patients With Hemophilic Arthropathy of the Knee and Ankle and Their Healthy Peers. A Case-control Study
Brief Title: Clinical, Functional and Musculoskeletal Differences Between Adult Patients With Hemophilia and Their Healthy Peers
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Investigación en Hemofilia y Fisioterapia (Network)
Responsible Party: Sponsor
Other Study IDs: He-BloodCC
Record Dates: First submitted 2022-10-18; First posted 2022-10-21 (Actual); Last update posted 2022-11-04 (Actual); Status verified 2022-11

CONDITIONS: Hemophilia Arthropathy
Keywords: Hemophilic arthropathy; Ankle; Knee; Strength; Muscle activation; Pressure pain threshold

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Hemophilia group: Patients with hemophilia, older than 18 years, with a diagnosis of hemophilic arthropathy of the knee and ankle. The different study variables will be evaluated following the indicated protocol.
  Interventions: Other: Clinical and functional assessment
- Healthy peers.group: Healthy subjects, older than 18 years, without joint damage at the time of the study, and physically active. The different study variables will be evaluated following the indicated protocol.
  Interventions: Other: Clinical and functional assessment

INTERVENTIONS:
Other: Clinical and functional assessment — The dependent variables (muscle strength, muscle activation, pressure pain threshold and joint status) and the outcome measures used to measure these variables will be: pressure dynamometer, surface electromyography, pressure algometer and Hemophilia Joint Health Score

SUMMARY:
Background. Hemophilia is characterized by the development of a progressive, degenerative, intra-articular lesion (hemophilic arthropathy). This arthropathy presents with chronic pain, limited range of motion, axial changes, and periarticular muscle atrophy.

Goal. To analyze the clonic, functional and musculoskeletal differences between adult patients with hemophilic arthropathy of the knee and ankle and their healthy peers.

Study design. Cases and controls study patients. 21 patients with hemophilia A and B and 21 subjects without joint damage.

Variables and measuring instruments: pressure pain threshold (pressure algometer); joint status (Hemophilia Joint Health Score scale); and strength (dynamometry) and muscle activation (surface electromyography).

Expected results. Observe the differences between patients with knee and ankle arthropathy and their healthy peers in muscle strength and activation.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with hemophilia A and B.
* Over 18 years
* With medical diagnosis of knee arthropathy
* With clinical evaluation by Hemophilia Joint Health Score
* In prophylactic treatment or on demand with FVIII / FIX concentrates for coagulation.
* Healthy subjects must meet knee joint health criteria; over 18 years; and no previous knee or ankle injuries in the 6 months prior to evaluation.

Exclusion Criteria:

* Patients with neurological or cognitive disorders that prevent the understanding of physical tests
* Not having signed the informed consent document

Ages: 18 Years to 45 Years | Sex: Male
Age Groups: Adult
Study Population: Patients with hemophilic arthropathy and their healthy pairs
Sampling Method: Non-Probability Sample
Enrollment: 42 (Estimated)
Dates: Start 2022-11-21 (Estimated); Primary Completion 2022-11-28 (Estimated); Study Completion 2022-12-23 (Estimated)

PRIMARY OUTCOMES:
Assess the muscle strength | Screening visit
  The force will be measured with a pressure dynamometer (Lafayette Manual muscle Tester model 01165). This device measures in Newton the force exerted by the patient in the requested muscular action. The higher the value, the greater muscle strength. We will perform the measurements bilaterally. Strength in the quadriceps and triceps surae muscles will be measured. The patient will be asked for 2 maximum isometric contractions of 5 seconds, with a rest of 30 seconds between them. In all the measurements, the evaluator will encourage the patient in a standardized way to carry out the contractions. In the measurement of the strength of all the muscles evaluated, the mean value of the measurements obtained will be used as a measure.

SECONDARY OUTCOMES:
Assess the muscle activation | Screening visit
  Muscle activation will be measured with surface electromyography (Shimmer Sensing model, Dublin, Ireland). Using this instrument, we will evaluate the electrical activity of the muscles and their level of activation. The placement of the electrodes will be marked on the subjects standing, and they will be placed following the European recommendations for the use of SEMG. A bipolar SEMG system will be used with circular electrodes 10 mm in diameter, 20 mm apart, placed longitudinally, in the direction of the muscle fibers studied, and with a reference electrode at a distance. The unit of measure is the μV. The higher the score, the greater muscle activation.
Assess the pressure pain threshold | Screening visit
  Pressure pain threshold will be measured with a pressure algometer (Wagner FPIXTM Digital Algometer model). This device measures in Newton/cm2 the pressure at which the subject perceives pressure pain. A pressure will be applied that we will increase at an approximate speed of 50kPa/s until the patient tells us that the sensation is beginning to be painful. In the knee we will measure bilaterally 3 cm medially to the midpoint of the inner edge of the patella, 2 cm proximally to the superior pole of the patella. At the ankle we will measure bilaterally ventrally to the lateral malleolus.
Assess the joint status | Screening visit
  In patients with hemophilia, joint status will be assessed with the Hemophilia Joint Health Score. This specific scale for use in patients with hemophilia is used to measure the joint status of patients with hemophilic arthropathy. It evaluates 8 items: inflammation and its duration, pain, muscle atrophy and strength, crackles, and loss of flexion and extension. It has a score of 0 (no joint damage) to 20 points (maximum joint damage) per joint (elbows, knees and ankles). A gait rating is added to 120 points (range 0-4 points), with the maximum rating on this scale being 124 points.

CONTACTS AND LOCATIONS:
Overall Officials: Rubén Cuesta-Barriuso, PhD, Principal Investigator — University of Oviedo

IPD SHARING:
Plan to Share IPD: No